CLINICAL TRIAL: NCT06865508
Title: Photo Biomodulation Therapy for Alveolar Osteitis Recovery in Oral Contraceptive Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Doaa Saeed Mohamed, Lecturer, Badr University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUC-IACUC-231015-38
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Alveolar Osteitis
Keywords: alveolar osteitis and oral contraceptive
MeSH Terms: conditions — Dry Socket | interventions — Laser Therapy

STUDY DESIGN:
Intervention Model Description: This study is a randomized clinical trial (RCT) designed to evaluate the effectiveness of laser therapy combined with zinc oxide eugenol dressing in comparison to zinc oxide eugenol dressing alone in the management of dry socket among females using oral contraceptives. The study assessed outcomes related to pain, quality of life, and socket volume.
Who Masked: Investigator, Outcomes Assessor
Masking Description: double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Experimental Group: Laser therapy combined with zinc oxide eugenol dressing. (Experimental): * Laser therapy was administered using a low-level laser device with the following parameters: [ wavelength 980 nm810, power 500mw, and duration 90 seconds (30second for each 3 sides].
  * Zinc oxide eugenol dressing was applied immediately before the laser therapy.
  * The intervention will be performed at [specified intervals every day 0, day7, day 14, day 30)]
  Interventions: Device: Laser therapy; Device: zinc oxide eugenol dressing.
- control group (Active Comparator): zinc oxide eugenol dressing.
  Interventions: Device: zinc oxide eugenol dressing.

INTERVENTIONS:
Device: Laser therapy — Laser therapy was administered using a low-level laser device with the following parameters: [ wavelength 980 nm810, power 500mw, and duration 90 seconds (30second for each 3 sides].
  Arms: 1. Experimental Group: Laser therapy combined with zinc oxide eugenol dressing.
Device: zinc oxide eugenol dressing. — zinc oxide eugenol dressing.

SUMMARY:
does laser effect on alveolar osteitis recovery in oral contraceptive users ?

DETAILED DESCRIPTION:
photo biomodulation therapy for alveolar osteitis recovery in oral contraceptive users

ELIGIBILITY:
* Inclusion Criteria:

Female patients aged 25-40 years. Currently using oral contraceptives for at least 3 months prior to participation.

Diagnosed with dry socket (alveolar osteitis) based on clinical criteria.

* Exclusion Criteria:

Presence of systemic diseases (e.g., diabetes, immunodeficiency disorders). Smoking or tobacco use. Allergies to zinc oxide or other study materials. Use of antibiotics or anti-inflammatory medications within the last 2 weeks. Pregnancy or breastfeeding.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
pain intensity by VAS | 4 weeks
  Pain intensity measured using a Visual Analog Scale (VAS) at day0, day7, day14 post-treatment.
Socket volume . | 4 weeks
  measured using [specific measurement technique, volumetric analysis] at day0, day14 and 1-month post-treatment

SECONDARY OUTCOMES:
Quality of life assessed | 4 weeks
  Quality of life assessed using the Oral Health Impact Profile (OHIP-5) questionnaire at day0, day7and day14 post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- physical therapy at Badr University in Cairo(BUC), Cairo, Egypt